CLINICAL TRIAL: NCT05698004
Title: A Wake Prone Positioning in Non-intubated Patients With Acute Hypoxemic Respiratory Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Montaser Gamal Ahmed (Other)
Responsible Party: Sponsor-Investigator, Montaser Gamal Ahmed, lecturer, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: prone positioning in ICU
Record Dates: First submitted 2022-12-30; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2022-12

CONDITIONS: Respiratory Failure, ICU
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Prone Position

STUDY DESIGN:
Intervention Model Description: Patients with acute hypoxemic respiratory failure attending the participating centres will receive either prone positioning + standard treatment or standard treatment only. All new acute hypoxemic respiratory failure patients will receive prone positioning + standard treatment for the first two weeks of the study. During the following two weeks, all new patients will receive standard treatment only. These cycles will be repeated until completion the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-1: prone positioning + standard treatment (Active Comparator): Patients randomized to the intervention group will be subjected to awake prone positioning. The target duration of prone positioning is 8 h/d to 10 h/d with 2 to 3 breaks (1-2 hours each), if needed. Daily prone positioning sessions will be protocolized to continue until 1 of the following stopping criteria is met: a relative improvement in the FIO2 requirement by 40% from the baseline value that sustained for 24 hours; endotracheal intubation; or discharge from the ICU. The treating team will supervise patients who could move themselves during the prone positioning process and assist the patients with positioning as required.
  Interventions: Other: prone positioning
- Group-2: Standard treatment only (No Intervention): Patients randomized to the control group, and their treating team, will be informed of their group assignment. Nurses instruct patients not to position themselves in the prone position.

INTERVENTIONS:
Other: prone positioning — The target duration of prone positioning is 8 h/d to 10 h/d with 2 to 3 breaks (1-2 hours each), if needed. Daily prone positioning sessions will be protocolized to continue until 1 of the following stopping criteria is met: a relative improvement in the FIO2 requirement by 40% from the baseline value that sustained for 24 hours; endotracheal intubation; or discharge from the ICU.
  Arms: Group-1: prone positioning + standard treatment

SUMMARY:
Patients admitted to the ICU with severe hypoxemia are at high risk for mortality. Few therapies have been proven to improve patient outcomes or duration of mechanical ventilation e.g. low tidal volume ventilation, prone positioning, and a fluid-restrictive strategy. Prone positioning is a technique used to help patients with acute respiratory distress syndrome breathe better. There is high degree of uncertainty on its effects on clinical outcomes in non-intubated patients with acute hypoxemia and larger studies are needed.

DETAILED DESCRIPTION:
we plan to study the effect of prone positioning versus standard treatment in non-intubated patients with acute hypoxemia admitted at Respiratory Intensive Care Unit (RICU), Chest Department, Assiut University Hospital, Egypt.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 years or older who are not intubated and required at least 40% oxygen (via low- or high-flow oxygen devices) or noninvasive positive pressure ventilation.

Exclusion Criteria: Patients will be excluded from the study if they :

had received invasive mechanical ventilation, had contraindications to prone positioning, are at risk of complications from prone positioning, had been self-prone positioning prior to enrollment and Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants within intervention arm whom need endotracheal intubation. | 30 days of randomization.
  Intubation is needed when one major criterion including (cardiac or respiratory arrest; hemodynamic instability, life threatening arrhythmias, inability to protect the airway; coma or psychomotor agitation and intolerance to NIV interface; and two of the following minor criteria: RR> 35/min., PaO2/FiO2<200 mmHg, and respiratory acidosis (pH<7.30)).

SECONDARY OUTCOMES:
Number of days on a ventilator. | 30 days of randomization.
  weaning considered successful if patient is able to achieve the following within 48 hours: pH >7.35, Decrease in PaCO2 of >15-20%, PaO2>60 mmHg, SaO2> 90% on FiO2 <40%, Respiratory rate < 24 bpm and No signs of respiratory distress like agitation, diaphoresis or anxiety.
mortality. | 60 days of randomization.
Length of ICU stay in days. | 60 days of randomization.
  duration of ICU stay from time of admission till discharge from ICU in days.
Length of hospital stay in days. | 60 days of randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Sahar Refaat Mahmoud, Principal Investigator — Assuit university hospital; Sarah Mohamed Hashem Hamza., Principal Investigator — Assuit university hospital; Emad Zareef, Principal Investigator — Assuit university hospital

REFERENCES:
- [Background] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337
- [Background] Matthay MA, Zemans RL, Zimmerman GA, Arabi YM, Beitler JR, Mercat A, Herridge M, Randolph AG, Calfee CS. Acute respiratory distress syndrome. Nat Rev Dis Primers. 2019 Mar 14;5(1):18. doi: 10.1038/s41572-019-0069-0. PMID 30872586
- [Background] Gattinoni L, Taccone P, Carlesso E, Marini JJ. Prone position in acute respiratory distress syndrome. Rationale, indications, and limits. Am J Respir Crit Care Med. 2013 Dec 1;188(11):1286-93. doi: 10.1164/rccm.201308-1532CI. PMID 24134414